CLINICAL TRIAL: NCT03189888
Title: Granulocyte-monocyte Apheresis in Steroid-dependent, Azathioprine-intolerant/Resistant Moderate Ulcerative Colitis: a Prospective Multicentre Study
Brief Title: Granulocyte-monocyte Apheresis in Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Arnaldo Amato, Principal Investigator, Valduce Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5/2012
Record Dates: First submitted 2017-06-13; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apheresis (Other): leukapheresis in ulcerative colitis
  Interventions: Device: apheresis

INTERVENTIONS:
Device: apheresis

SUMMARY:
BACKGROUND: Granulocyte-monocyte apheresis has been proposed for the treatment of ulcerative colitis, although is limited by costs and variability of results.

ELIGIBILITY:
Inclusion Criteria:

* moderate UC with steroid-dependence and azathioprine intolerance or resistance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
steroid-free clinical remission | 3 months

REFERENCES:
- [Derived] Imperiali G, Amato A, Terpin MM, Beverina I, Bortoli A, Devani M, Vigano C; Study Group on IBD (GSMII). Granulocyte-Monocyte Apheresis in Steroid-Dependent, Azathioprine-Intolerant/Resistant Moderate Ulcerative Colitis: A Prospective Multicenter Study. Gastroenterol Res Pract. 2017;2017:9728324. doi: 10.1155/2017/9728324. Epub 2017 Dec 21. PMID 29403531